CLINICAL TRIAL: NCT00798096
Title: Phase II, Multicenter, Simon Two-Stage Study of Fostamatinib Disodium in Patients With Relapsed or Refractory T-Cell Lymphoma
Brief Title: Efficacy and Safety Study of Fostamatinib Disodium Tablets to Treat T-Cell Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Rigel Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D4300C00024; C-935788-017 (Other: Rigel Pharmaceuticals)
Record Dates: First submitted 2008-11-21; First posted 2008-11-25 (Estimated); Results first posted 2014-06-12 (Estimated); Last update posted 2016-09-19 (Estimated); Status verified 2016-08

CONDITIONS: T Cell Lymphoma
Keywords: T Cell Lymphoma; Lymphoma
MeSH Terms: conditions — Lymphoma, T-Cell; Lymphoma | interventions — fostamatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Fostamatinib Disodium

INTERVENTIONS:
Drug: Fostamatinib Disodium — 200 mg PO BID
  Other Names: Code Designation: R935788 Sodium Hexahydrate; USAN Name: Fostamatinib Disodium; CAS No.: 914295-16-2

SUMMARY:
Patients meeting specific inclusion and exclusion criteria will be enrolled in two stages, 19 patients in Stage 1 and 36 patients in Stage 2. Stage 2 will enroll if 4 or more patients exhibit a response at Week 8 or later in the study. All enrolled patients will be treated with Fostamatinib Disodium until disease progression. Efficacy will be assessed by tumor measurements using CT and PET (when indicated) scans and physical exam at baseline, and scans and physical exam of all disease-involved areas every 8 weeks until progression. Safety will be assessed by periodic physical exams, clinical laboratory studies, and adverse events. All patients will have a follow-up visit 30 days following last study drug treatment. Blood samples for PK assessment will be obtained from all patients enrolled in Stage 1 at protocol defined intervals.

DETAILED DESCRIPTION:
Up to 61 patients (male and female) meeting the inclusion and exclusion criteria will be enrolled into this trial in two stages. All enrolled patients will be treated with R788 at 200 mg PO bid until disease progression. In the initial stage of the study, a total of 19 patients will be enrolled and treated with Fostamatinib Disodium. Should at least 4 patients exhibit a response at Week 8 or later of the study, the second stage of 36 patients will open to enrollment. Efficacy will be assessed by CT and PET scans (when indicated) and physical exam at baseline, and CT scans and physical exam of all disease-involved areas every 8 weeks until progression. Safety will be assessed by periodic physical exams, clinical laboratory studies, and adverse events. All patients will have a follow-up visit 30 days following last study drug treatment. Blood samples for PK assessment will be obtained from all patients enrolled in Stage 1 at protocol-defined intervals. Patients with accessible tumor tissue will be asked to undergo a biopsy for a fresh tissue sample for assessment of Syk activity in tumor tissue. Archived tissue samples from the initial diagnostic biopsy and the most recent biopsy for lymphoma will be obtained in the event a fresh tumor biopsy cannot be obtained. Patients who have accessible tumor tissue will be asked to consent to a second tumor biopsy at Week 8, to assess the impact of Fostamatinib Disodium treatment on the activity of Syk and its downstream markers. All baseline fresh or archived tumor tissue samples will undergo central pathology review to confirm the diagnosis of TCL.

ELIGIBILITY:
Inclusion Criteria:

* Patients must give written informed consent to participate in this study by signing an IRB/EC-approved Informed Consent Form (ICF) prior to admission to this study.
* Males and females, 18 years of age or older.
* Patients must have histologically proven T-cell lymphoma (TCL).
* Patients must have documented disease progression after receiving at least one prior therapeutic regimen and must be patients for whom no known curative therapy exists.

Exclusion Criteria:

* Patient has a history of, or a concurrent, clinically significant illness, medical condition or laboratory abnormality that, in the investigator's opinion, could affect the conduct of the study.
* Has a B-cell lymphoma, primary CNS lymphoma, or known lymphomatous involvement of the CNS, or any other NK/T-cell leukemia/lymphoma.
* Has uncontrolled or poorly controlled hypertension.
* Has had recent (within 1 month prior to Day 1) serious surgery or uncontrolled infectious disease.
* Has any concurrent malignancy requiring treatment.
* Has a known positive test for Hepatitis B surface Ag, Hepatitis C, or HIV.
* Has laboratory abnormalities.
* Has difficulty swallowing or malabsorption.
* Has an ECOG performance status > 2.
* Has not recovered from adverse effects related to last prior therapy for lymphoma.
* Has had an allotransplantation within 90 days prior to Day 1 of treatment.
* Has been treated with a CYP3A4 inducer/inhibitor within 3 days prior to Day 1 of treatment or is expected to require treatment with CYP3A4 inducer/inhibitor during the course of the study.
* Has received systemic steroids at a dose greater than the equivalent of 10 mg/day of prednisone within 7 days prior to Day 1 of treatment.
* Has received any other investigational therapy within 5 half-lives of the agent or 2 weeks of Day 1 of treatment, whichever is longer.
* Is a female of childbearing potential unless menopausal, surgically sterile, or willing to use an effective method of birth control, (oral contraceptive, mechanical barrier, long-acting hormonal agent), during the study and for 30 days thereafter.
* Is pregnant or lactating.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2009-03; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Skolnik, MD, Study Director — AstraZeneca
Locations (10):
- United States (8):
  - Research Site, San Francisco, California
  - Research Site, Stanford, California
  - Research Site, Atlanta, Georgia
  - Research Site, Boston, Massachusetts
  - Research Site, Rochester, Minnesota
  - Research Site, Omaha, Nebraska
  - Research Site, New York, New York
  - Research Site, Houston, Texas
- Canada (2):
  - Research Site, Vancouver, British Columbia
  - Research Site, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: D4300C00024 Clinical Study Report — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_6111&studyid=1482&filename=D4300C00024_C935788-017.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 18 patients with T-Cell lymphoid malignancy were enrolled in this study from 05 March 2009 until 04 January 2010. As of 19 May 2010, no patients remain on study. All enrolled patients received at least one dose of fostamatinib. This study was conducted at 9 sites in the U.S. and Canada.
Pre-assignment Details: There was a screening period of up to 28 days, after which if all inclusion/exclusion criteria were met, patients were dosed with fostamatinib treatment for a treatment period of 8 weeks. Patients could continue treatment until disease progression, toxicity or withdrawal from the study
Groups:
- Overall Study: 1-fostamatinib 200mg, BID, Oral
Period: Overall Study
Arm/Group | Overall Study
Started | 18 (Treatment with 200 mg bid, oral Fostamatanib until disease progression, toxicity or withdrawal)
Completed | 16 (Completion of Study is defined as a minimum of 8 weeks of treatment or early disease progression)
Not Completed | 2
Not completed — Ongoing | 2

BASELINE CHARACTERISTICS:
Arm/Group | Overall Study
Number analyzed (Participants) | 18
Age, Continuous [Mean (Standard Deviation); unit: Years] | 68.5 (12) [44 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 10
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian | 2
  White | 15
  Other - Unknown | 1

OUTCOME MEASURES:

1. Primary Outcome: The Primary Efficacy Endpoint for This Study is Overall Regressive Response Rate (ORRR): Proportion of Patients With a Best Response of Complete Response (CR), Partial Response (PR), or Regressive Stable Disease (RSD).
Description: Overall regressive response rate (ORRR) is the proportion of patients with a best response of Complete Response (CR), Partial Response (PR) (per Cheson 2007), or Regressive Stable Disease (RSD) defined as regressive disease that does not meet the criteria for partial response.
Time Frame: Serial tumor assessments were taken at baseline (within 28 days of the start of treatment), and re-evaluated at Day 57, and every 8weeks therafter or to confirm response . (Maximum duration of treatment 182 days, Maximum duration of follow-up 217 days)
Measure: Number; unit: Participants
Arm/Group | Overall Study
Number analyzed (Participants) | 18
Participants | 4

2. Secondary Outcome: Clinical Benefit Rate is the Proportion of Patients With Best Response of Complete Response (CR), Partial Response (PR), or Stable Disease (SD).
Description: Clinical benefit rate is the proportion of patients with best response of Complete Response (CR), Partial Response (PR), or Stable Disease (SD).
Time Frame: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Overall Study
Number analyzed (Participants) | 18
Participants | 5

3. Secondary Outcome: Overall Response Rate (ORR) is the Proportion of Patients With a Best Response of Complete Response (CR) or Partial Response (PR).
Description: Overall response rate (ORR) is the proportion of patients with a best response of Complete Response (CR) or Partial Response (PR).
Time Frame: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Overall Study
Number analyzed (Participants) | 18
Participants | 0

4. Secondary Outcome: Duration of Overall Response is the Time From First Documentation of Complete or Partial Response, Whichever Occurs Earlier, to Discontinuation of Study Drug.
Description: Duration of Overall Response is the time from first documentation of Complete or Partial Response (Cheson 2007), whichever occurs earlier, to discontinuation of study drug.
Time Frame: as for outcome 1
Measure: Median (Standard Deviation); unit: Days
Arm/Group | Overall Study
Number analyzed (Participants) | 18
Days | NA (NA) [NA to NA] — Duration of response could not be calculated since 0 patients responded.

ADVERSE EVENTS:
Arm/Group | Overall Study
Serious Adverse Events (participants affected / at risk) | 11/18
Other Adverse Events (participants affected / at risk) | 18/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Overall Study (N=18)
Febrile Neutropenia (Blood and lymphatic system disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Melaena (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 2
Pyrexia (General disorders) | 1
Hepatic Failure (Hepatobiliary disorders) | 1
Lobar Pneumonia (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Sepsis (Infections and infestations) | 2
Skin Infection (Infections and infestations) | 1
Wound Secretion (Injury, poisoning and procedural complications) | 1
Anorexia (Metabolism and nutrition disorders) | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Overall Study (N=18)
Anaemia (Blood and lymphatic system disorders) | 3
Febrile Neutropenia (Blood and lymphatic system disorders) | 2
Neutropenia (Blood and lymphatic system disorders) | 7
Pancytopenia (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 7
Tachycardia (Cardiac disorders) | 3
Inappropriate Antidiuretic Hormone Secretion (Endocrine disorders) | 1
Eye Irritation (Eye disorders) | 1
Eye Pain (Eye disorders) | 1
Lacrimation Increased (Eye disorders) | 2
Vision Blurred (Eye disorders) | 2
Abdominal Distension (Gastrointestinal disorders) | 2
Abdominal Pain (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 3
Defaecation Urgency (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 7
Dry Mouth (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Flatulence (Gastrointestinal disorders) | 1
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 1
Gingival Bleeding (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 7
Oral Mucosal Blistering (Gastrointestinal disorders) | 1
Oral Pain (Gastrointestinal disorders) | 1
Rectal Haemorrhage (Gastrointestinal disorders) | 1
Stomatitis (Gastrointestinal disorders) | 2
Tongue Ulceration (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 7
Asthenia (General disorders) | 1
Chest Pain (General disorders) | 1
Chills (General disorders) | 7
Face Oedema (General disorders) | 3
Fatigue (General disorders) | 11
Localised Oedema (General disorders) | 1
Mucosal Inflammation (General disorders) | 2
Oedema (General disorders) | 1
Oedema Peripheral (General disorders) | 4
Pain (General disorders) | 1
Pyrexia (General disorders) | 8
Hyperbilirubinaemia (Hepatobiliary disorders) | 2
Candidiasis (Infections and infestations) | 1
Central Line Infection (Infections and infestations) | 1
Cystitis (Infections and infestations) | 1
Fungal Infection (Infections and infestations) | 1
Fungal Skin Infection (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Nail Infection (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 2
Skin Infection (Infections and infestations) | 1
Upper Respiratory Tract Infection (Infections and infestations) | 2
Urinary Tract Infection (Infections and infestations) | 2
Urinary Tract Infection Bacterial (Infections and infestations) | 1
Wound Infection (Infections and infestations) | 1
Wound Secretion (Injury, poisoning and procedural complications) | 1
Alanine Aminotransferase Increased (Injury, poisoning and procedural complications) | 1
Aspartate Aminotransferase Increased (Injury, poisoning and procedural complications) | 6
Blood Albumin Decreased (Injury, poisoning and procedural complications) | 1
Blood Alkaline Phosphatase Increased (Injury, poisoning and procedural complications) | 2
Blood Bicarbonate Decreased (Injury, poisoning and procedural complications) | 1
Blood Bilirubin Increased (Injury, poisoning and procedural complications) | 1
Blood Creatine Increased (Injury, poisoning and procedural complications) | 1
Blood Glucose Increased (Injury, poisoning and procedural complications) | 1
Blood Lactate Dehydrogenase Increased (Injury, poisoning and procedural complications) | 1
Blood Magnesium Decreased (Injury, poisoning and procedural complications) | 1
Blood Phosphorus Decreased (Injury, poisoning and procedural complications) | 1
Blood Potassium Decreased (Injury, poisoning and procedural complications) | 1
Blood Potassium Increased (Injury, poisoning and procedural complications) | 1
Blood Sodium Decreased (Injury, poisoning and procedural complications) | 1
Blood Sodium Increased (Injury, poisoning and procedural complications) | 1
Haemoglobin Decreased (Injury, poisoning and procedural complications) | 4
Platelet Count Decreased (Injury, poisoning and procedural complications) | 1
Urine Output Decreased (Injury, poisoning and procedural complications) | 1
Weight Decreased (Injury, poisoning and procedural complications) | 1
White Blood Cell Count Decreased (Injury, poisoning and procedural complications) | 2
White Blood Cell Count Decreased (Injury, poisoning and procedural complications) | 5
Decreased Appetite (Metabolism and nutrition disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 2
Hypercalcaemia (Metabolism and nutrition disorders) | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 4
Hypophosphataemia (Metabolism and nutrition disorders) | 1
Hypovolaemia (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 2
Bone Pain (Musculoskeletal and connective tissue disorders) | 1
Buttock Pain (Musculoskeletal and connective tissue disorders) | 1
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 1
Neck Pain (Musculoskeletal and connective tissue disorders) | 1
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 2
Shoulder Pain (Musculoskeletal and connective tissue disorders) | 2
Dizziness (Nervous system disorders) | 5
Dysgeusia (Nervous system disorders) | 2
Headache (Nervous system disorders) | 5
Memory Impairment (Nervous system disorders) | 1
Neuropathy Peripheral (Nervous system disorders) | 1
Parosmia (Nervous system disorders) | 1
Peripheral Sensory Neuropathy (Nervous system disorders) | 2
Poor Quality Sleep (Nervous system disorders) | 1
Sinus Headache (Nervous system disorders) | 1
Depression (Psychiatric disorders) | 1
Hallucination (Psychiatric disorders) | 1
Dysuria (Renal and urinary disorders) | 1
Pollakiuria (Renal and urinary disorders) | 1
Renal Failure Acute (Renal and urinary disorders) | 1
Oedema Genital (Reproductive system and breast disorders) | 1
Apnoea (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 5
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 1
Nasal Dryness (Respiratory, thoracic and mediastinal disorders) | 1
Pharyngolaryngeal Pain (Respiratory, thoracic and mediastinal disorders) | 2
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1
Upper Respiratory Tract Congestion (Respiratory, thoracic and mediastinal disorders) | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 1
Erythema (Skin and subcutaneous tissue disorders) | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 3
Night Sweats (Skin and subcutaneous tissue disorders) | 2
Pain Of Skin (Skin and subcutaneous tissue disorders) | 1
Periorbital Oedema (Skin and subcutaneous tissue disorders) | 2
Rash (Skin and subcutaneous tissue disorders) | 1
Rash Erythematous (Skin and subcutaneous tissue disorders) | 1
Skin Disorder (Skin and subcutaneous tissue disorders) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1
Haematoma (Vascular disorders) | 1
Hot Flush (Vascular disorders) | 1
Hypertension (Vascular disorders) | 4

LIMITATIONS AND CAVEATS:
This is a small, non-randomized study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
An Investigator agrees to provide a copy of the publication to AstraZeneca for review at least 30 days in advance of submission for publication. Investigators in multicenter (MC) studies agree to postpone MC publications until the earlier of the date of the first AstraZeneca authorized MC publication or a period up to 18 months from study completi